CLINICAL TRIAL: NCT05969522
Title: Stratified Therapy on Pediatric AAGN Based on Risk Assessment-A Prospective, Multicenter, Open, Tendentious Matched Control Clinical Study
Brief Title: Stratified Therapy on Pediatric AAGN
Acronym: STPARS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wang Mo (Other)
Responsible Party: Sponsor-Investigator, Wang Mo, Professor/Chief Physician, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ANCA20230706
Record Dates: First submitted 2023-07-10; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis; ANCA-Associated Glomerulonephritis
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Glucocorticoids; Rituximab; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group-Low and medium risk group (Other): The children with AAGN admitted to all cooperating units during 2017.01.01 to 2022.12.31 were followed up for more than 6 months, and the case data were complete.
  PARRG Classification (pediatric AAGN renal risk grade, pediatric AAV renal risk grade, PARRG) According to the PARRG grading method provided by the Affiliated Children's Hospital of Chongqing Medical University, the enrolled children with AAGN were classified into high risk group, medium risk group, low risk group, medium risk group, low risk combination and low risk group according to the two indexes of eGFR and percentage of glomerular sclerosis during renal biopsy.
  PARRG risk grading criteria:
  There are two risk factors for ESRD: (1) eGFR≤20ml/min/1.73m2 at renal biopsy; ② The proportion of glomerular sclerosis ≥30%; High risk resistance: meet 2 risk factors; Moderate risk group: only 1 risk factor; Low risk group: no above risk factors;
  Interventions: Drug: GlucoCorticoid
- Control group-High risk group (Other): The children with AAGN admitted to all cooperating units during 2017.01.01 to 2022.12.31 were followed up for more than 6 months, and the case data were complete.
  PARRG Classification (pediatric AAGN renal risk grade, pediatric AAV renal risk grade, PARRG) According to the PARRG grading method provided by the Affiliated Children's Hospital of Chongqing Medical University, the enrolled children with AAGN were classified into high risk group, medium risk group, low risk group, medium risk group, low risk combination and low risk group according to the two indexes of eGFR and percentage of glomerular sclerosis during renal biopsy.
  PARRG risk grading criteria:
  There are two risk factors for ESRD: (1) eGFR≤20ml/min/1.73m2 at renal biopsy; ② The proportion of glomerular sclerosis ≥30%; High risk resistance: meet 2 risk factors; Moderate risk group: only 1 risk factor; Low risk group: no above risk factors;
  Interventions: Drug: GlucoCorticoid
- Experimental group-Low and medium risk group (Experimental): Newly diagnosed children with AAGN admitted to our partners during the period of 2023.01.01 to 2023.12.31.
  All children with AAGN were PARRG risk graded before treatment with RTX and CTX:
  PARRG Classification (pediatric AAGN renal risk grade, pediatric AAV renal risk grade, PARRG) According to the PARRG grading method provided by the Affiliated Children's Hospital of Chongqing Medical University, the enrolled children with AAGN were classified into high risk group, medium risk group, low risk group, medium risk group, low risk combination and low risk group according to the two indexes of eGFR and percentage of glomerular sclerosis during renal biopsy.
  PARRG risk grading criteria:
  There are two risk factors for ESRD: (1) eGFR≤20ml/min/1.73m2 at renal biopsy; ② The proportion of glomerular sclerosis ≥30%; High risk resistance: meet 2 risk factors; Moderate risk group: only 1 risk factor; Low risk group: no above risk factors;
  Interventions: Drug: GlucoCorticoid
- Experimental group-High risk group (Experimental): Newly diagnosed children with AAGN admitted to our partners during the period of 2023.01.01 to 2023.12.31.
  All children with AAGN were PARRG risk graded before treatment with RTX and CTX:
  PARRG Classification (pediatric AAGN renal risk grade, pediatric AAV renal risk grade, PARRG) According to the PARRG grading method provided by the Affiliated Children's Hospital of Chongqing Medical University, the enrolled children with AAGN were classified into high risk group, medium risk group, low risk group, medium risk group, low risk combination and low risk group according to the two indexes of eGFR and percentage of glomerular sclerosis during renal biopsy.
  PARRG risk grading criteria:
  There are two risk factors for ESRD: (1) eGFR≤20ml/min/1.73m2 at renal biopsy; ② The proportion of glomerular sclerosis ≥30%; High risk resistance: meet 2 risk factors; Moderate risk group: only 1 risk factor; Low risk group: no above risk factors;
  Interventions: Drug: GlucoCorticoid

INTERVENTIONS:
Drug: GlucoCorticoid — The high-risk group: methylprednisolone intravenous 15-30mg/kg/d (Max.500mg/d)*3 days , with 2 courses, interval 5-7 days;Oral prednisone acetate 1.5-2mg/kg/d (Max. 60mg/d) during methylprednisolone impact interval and later stage, with the first reduction after 2-4 weeks. The dose was reduced once every 3 weeks in the first 3 months, and once every 4 weeks in the next 3 months, with a reduction of 5-10mg/ day each time; Rituximab：375 mg/m2/ time, once a week for 4 times;Intravenous cyclophosphamide 7.5-10mg/kg.d*2 days(Max.500mg/d), once every 4 weeks, twice in total, at the 8th and 12th week.The medium-low risk group: methylprednisolone was the same dose as before, but only with 1 course, then followed by oral prednisone acetate 1.5-2mg/kg/d (Max. 60mg/d), divided into three times for 3 weeks, and then changed to morning daily; The dose was reduced as the high-risk group ;Rituximab was the same dose as before.
  Other Names: Rituximab; Cyclophosphamide

SUMMARY:
Clinical information of children with ANCA-associated nephritis admitted to Children's Hospital Affiliated to Chongqing Medical University and partner centers from January 1, 2023 to December 31, 2023 was collected:

To evaluate and compare the differences in survival, renal outcomes, and adverse reactions in children with ANCA-associated nephritis given different interventions according to the revised PARRG risk stratification, and to evaluate the superiority of ANCA-associated nephritis given according to the revised PARRG risk stratification.

(2) To evaluate the efficacy and safety of glucocorticoid combined with rituximab and cyclophosphamide as induction regimen in high-risk group and glucocorticoid combined with rituximab as induction regimen in children with ANCA-associated nephritis (AAGN) in low and middle risk group based on PARRG risk stratification

ELIGIBILITY:
Inclusion Criteria:

* 1) Newly diagnosed AAGN patients with onset age of 5-17 years, complete renal biopsy and regular follow-up in the hospital; 2) All enrolled children met the following inclusion criteria: ANCA classification criteria: Patients who meet the 2007 European Medicines Agency (EMA) classification algorithm or the 2012 CHCC definition. Clinical classification includes: micropolyvasculitis (MPA), granulomatous polyvasculitis (GPA) and eosinophilic granulomatous polyvasculitis (EGPA);

AAGN diagnostic criteria: ANCA vasculitis combined with any of the following:

1. Hematuria: gross hematuria or microscopic hematuria: 3 times microscopic hematuria within 1 week: red blood cells &gt in urine routine; 3 / high magnification field (HP) or > 17 /ul (higher than normal value, can be adjusted according to the standard of the laboratory of each center);
2. proteinuria: meet any of the following: ① 3 times in 1 week urine routine protein positive; 2) 24h urinary protein quantification > 150 mg or urinary protein/creatinine (mg/mg)> 0.2; 3 urinary microalbumin higher than normal for 3 times in 1 week;
3. Renal insufficiency: increased serum creatinine > 10% base or decreased creatinine clearance > 25%.

Exclusion Criteria:

- 1) Patients who relied on dialysis for more than 1 month at the time of diagnosis, or the proportion of glomerular sclerosis ≥75% at the time of renal biopsy; 2) Patients with severe infection (such as diffuse peritonitis, severe pneumonia, cellulitis, active Epstein-Barr virus infection, active cytomegalovirus infection, hepatitis B virus infection, tuberculosis infection, fungal infection, etc.) and tumor.

3) Patients with other primary or secondary kidney diseases (such as IgA nephropathy, membranous nephropathy, anti-glomerular basement membrane nephritis, polycystic kidney disease, renal dysplasia, urinary tract malformation, etc.); 4) Parents or children refused to join the group.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate (complete and partial response rate) | 6 months
  The rate of complete or partial response to ANCA vasculitis-associated nephritis (AAGN) was assessed at 6 months. Complete AAGN response was defined as: 1. Estimated glomerular filtration rate (eGFR) ≥60ml/min/1.73m2, or a decrease of less than 15% from baseline eGFR; 2. Proteinuria ≤0.3g/24 hours.Partial AAGN response was defined as: 1. Estimated glomerular filtration rate (eGFR) ≥30ml/min/1.73m2, or a reduction of less than 50% from baseline eGFR; 2. Decreased proteinuria>Baseline 50% or 24-hour urinary protein quantification<50mg/Kg.d.

SECONDARY OUTCOMES:
The time to achieve complete and partial AAGN remission | 6 months
  The time to achieve complete and partial AAGN remission

CONTACTS AND LOCATIONS:
Overall Officials: mo Wang, Study Director — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China